CLINICAL TRIAL: NCT01469000
Title: A Randomised Phase 2 Trial of Pemetrexed and Gefitinib Versus Gefitinib as First Line Treatment for Patients With Stage IV Non-Squamous Non-Small Cell Lung Cancer With Activating Epidermal Growth Factor Receptor Mutations
Brief Title: A Study of Pemetrexed and Gefitinib Versus Gefitinib in Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14034; H3E-CR-JMIT (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Results first posted 2016-04-28 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Carcinoma, Non Small Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 250 mg Gefitinib/500 mg Pemetrexed (Experimental): 250 milligrams (mg) Gefitinib taken orally once daily (QD) and 500 milligrams per square meter (mg/m²) Pemetrexed taken intravenously (IV) once every 3 weeks concurrently with Gefitinib taken orally QD.
  Interventions: Drug: Gefitinib; Drug: Pemetrexed
- 250 mg Gefitinib (Active Comparator): 250 milligrams (mg) Gefitinib taken orally QD
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — 250 mg orally once per day. Number of cycles until disease progression or unacceptable toxicity develops.
  Other Names: Iressa
Drug: Pemetrexed — 500 mg/m² IV on day 1 of each 21 day cycle. Number of cycles until disease progression or unacceptable toxicity develops.
  Other Names: Alimta
  Arms: 250 mg Gefitinib/500 mg Pemetrexed

SUMMARY:
The purpose of this study is to compare the combination of pemetrexed and gefitinib versus gefitinib alone, in terms of progression-free survival. This study is in participants who have stage IV non squamous NSCLC with activating epidermal growth factor mutations and who have not had any previous chemotherapy for stage IV disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced (Stage IV) or recurrent non-squamous NSCLC
* Eligible participants of reproductive potential must agree to use adequate contraceptive methods during the study period and for at least 6 months after the last dose of study therapy
* Negative pregnancy test for women of childbearing potential
* Males or females, aged 18 years or above
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* The participant's primary NSCLC tumor has an activating Epidermal Growth Factor Receptor (EGFR) mutation, as determined by any validated method
* The participant consents to provide a tissue sample for prestudy EGFR mutation testing and the tumor tissue sample is available for detection of EGFR expression and other markers for centralized testing by Lilly
* The participant has measurable disease at the time of study entry, documented by computed tomography (CT) scan or magnetic resonance imaging (MRI), as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* The participant has not had any prior systemic chemotherapy, immunotherapy, or biological therapy (for example, targeted therapy, such as erlotinib or gefitinib) for Stage IV or recurrent non-squamous NSCLC
* The participant has adequate organ function, defined as:

  * White blood cell count ≥3 x 10^9/liter (L); absolute neutrophil count (segmented and bands) ≥1.5 x 10^9/L; platelet count ≥100 x 10^9/L; hemoglobin ≥9.0 gram per deciliter (g/dL)
  * Total bilirubin ≤1.5 times the upper limit of the normal (ULN) range; and alkaline phosphatase (AP), aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 times ULN (or ≤5 times ULN if the liver has tumor involvement)
  * Calculated creatinine clearance ≥45 milliliter per minute (mL/min)
* The participant is able to take folic acid, vitamin B12, and dexamethasone, according to the protocol's requirements
* Life expectancy of at least 3 months
* Provision of informed consent
* Prior radiation therapy is allowed to <25% of the bone marrow; however, prior radiation to the whole pelvis not allowed. Prior radiation therapy must be completed at least 2 weeks prior to first study-drug administration. Participants must have recovered from the acute toxic effects prior to first study-drug administration.

Exclusion Criteria:

* The participant has received prior chemotherapy for advanced and/or metastatic disease, or adjuvant/neoadjuvant treatment with pemetrexed or an EGFR-tyrosine Kinase inhibitor (TKI)
* The participant's tumor contains predominantly small cell lung cancer or squamous NSCLC
* The participant is receiving concurrent treatment with any other anticancer therapy, including other chemotherapy, immunotherapy, hormonal therapy, chemoembolization, biological or targeted therapy, or radiotherapy (palliative irradiation of bone lesions is allowed)
* The participant has untreated central nervous system (CNS) metastases Participants with treated brain metastases are eligible if they are clinically stable with regard to neurologic function, off steroids after cranial irradiation (whole brain radiation therapy, focal radiation therapy, stereotactic radiosurgery) ending at least 2 weeks before enrollment, or after surgical resection performed at least 28 days before enrollment. No evidence of Grade ≥1 CNS hemorrhage based on pretreatment MRI or Intravenous (IV) contrast CT scan (performed within 21 days before randomization).
* The participant has undergone radiotherapy within 28 days before enrollment (localized radiotherapy for pain relief allowed, provided 25% or less of their total bone marrow had been irradiated)
* The participant has clinically relevant congestive heart failure (New York Heart Association [NYHA] II-IV) or symptomatic or poorly controlled cardiac arrhythmia
* The participant has a serious illness or medical condition that would compromise their safety or impair their ability to comply with the protocol's requirements, including, but not limited to, the following:

  * Known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)-related illness
  * Active or uncontrolled clinically serious infection
  * Previous or concurrent malignancy except for basal or squamous cell skin cancer and/or in situ carcinoma of the cervix, or other solid tumors treated curatively and without evidence of recurrence for at least 5 years prior to the study
  * Uncontrolled metabolic disorders or other nonmalignant organ or systemic diseases or secondary effects of cancer that induce a high medical risk and/or make assessment of survival uncertain
  * Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the participant ineligible for entry into this study
  * The participant has significant third space fluid retention, and is not amenable for required repeated drainage
  * Known allergy or hypersensitivity reaction to any of the treatment components
* Are unable to interrupt aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs), other than an aspirin dose ≤1.3 grams per day, for at least 2 days (5 days for long-acting agents [for example, piroxicam]) before, during, and for at least 2 days after administration of pemetrexed
* Concomitant use of cytochrome P450 (CYP)3A4 inducers or CYP3A4 inhibitors
* Participants under therapy with warfarin or coumarin derivatives who are unable to switch to low molecular weight heparin, unless regular monitoring of changes in prothrombin time (PT) (PT/international normalized ratio [INR]) will be applicable
* Any known significant ophthalmologic abnormalities of the surface of the eye. The use of contact lenses is not recommended during the study
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or non-approved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study Participants participating in surveys or observational studies are eligible to participate in this study
* The participant has previously received treatment with gefitinib, erlotinib or pemetrexed
* Any evidence of clinically active interstitial lung disease. Asymptomatic participants with chronic, stable, radiographic changes are eligible.
* Have preexisting idiopathic pulmonary fibrosis as evidenced by computed tomography (CT) scan/x-ray at baseline; have or had any disease of acute lung injury, idiopathic pulmonary fibrosis, pulmonary pneumonia, or pneumoconiosis evident on an x-ray; have or had any disease of radiation pneumonia or drug-induced pneumonia, which requires treatment with corticosteroids.
* The participant is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2012-02; Primary Completion 2015-04 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (25):
- China (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changchun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changsha
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sichuan
- Japan (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamaguchi
- South Korea (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cheong Ju-City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
- Taiwan (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Keelung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuei Shan Hsiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niao Sung Hsiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zhonghe

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Cheng Y, Murakami H, Yang PC, He J, Nakagawa K, Kang JH, Kim JH, Wang X, Enatsu S, Puri T, Orlando M, Yang JC. Randomized Phase II Trial of Gefitinib With and Without Pemetrexed as First-Line Therapy in Patients With Advanced Nonsquamous Non-Small-Cell Lung Cancer With Activating Epidermal Growth Factor Receptor Mutations. J Clin Oncol. 2016 Sep 20;34(27):3258-66. doi: 10.1200/JCO.2016.66.9218. Epub 2016 Aug 9. PMID 27507876

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who were alive and completed the follow-up period or who died were considered to have completed the study.
Groups:
- 250 mg Gefitinib/500 mg Pemetrexed: 250 milligrams (mg) Gefitinib taken orally once daily (QD) and 500 milligrams per square meter (mg/m²) Pemetrexed taken intravenously (IV) once every 3 weeks concurrently with Gefitinib QD.
- 250 mg Gefitinib: 250 mg Gefitinib taken orally once QD
Period: Overall Study
Arm/Group | 250 mg Gefitinib/500 mg Pemetrexed | 250 mg Gefitinib
Started | 129 | 66
Received at Least 1 Dose of Study Drug | 126 | 65
Completed | 109 | 62
Not Completed | 20 | 4
Not completed — Withdrawal by Subject | 16 | 3
Not completed — Sponsor Decision | 4 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 250 mg Gefitinib/500 mg Pemetrexed | 250 mg Gefitinib | Total
Number analyzed (Participants) | 126 | 65 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.11 (9.36) | 60.94 (9.45) | 61.71 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 41 | 123
  Male | 44 | 24 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 126 | 65 | 191
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 126 | 65 | 191
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 33 | 19 | 52
  Japan | 42 | 15 | 57
  Taiwan | 28 | 13 | 41
  Korea, Republic of | 23 | 18 | 41

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization to the first date of objectively determined progressive disease or death from any cause,whichever is earlier.The censoring is taken in the following order: If a participant didn't have a complete baseline disease assessment,then the PFS time was censored at the enrollment date, regardless of whether or not objectively determined disease progression or death has been observed for the participant;otherwise,if a participant is not known to have died or have objective progression as of the data inclusion cutoff date for the analysis,the PFS time will be censored at the last complete objective progression-free disease assessment date.Progressive disease (PD) was defined as at least a 20% increase in the sum of the diameters of target lesions,taking as reference the smallest sum on study. Also,the sum must also demonstrate an absolute increase of at least 5 millimeter (mm).The appearance of one or more new lesions is also considered progression.
Time Frame: Randomization to Progressive Disease or Death Due to Any Cause (Up to 58.78 Months)
Population: All participants who received at least 1 dose of study drug. Participants censored: Gefitinib/Pemetrexed =24, Gefitinib=3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 250 mg Gefitinib/500 mg Pemetrexed | 250 mg Gefitinib
Number analyzed (Participants) | 126 | 65
Months | 16.23 [12.58 to 18.73] | 11.07 [9.66 to 13.83]
Statistical Analysis 1: Comparison: 250 mg Gefitinib/500 mg Pemetrexed vs 250 mg Gefitinib; Test type: Superiority or Other; p = 0.009, Regression, Cox — 1-sided; Adjusted for gender, performance status, previous adjuvant /neoadjuvant treatment, age, smoking history, mutation type, and country; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.48 to 0.93]

2. Secondary Outcome: Time To Progressive Disease (TTPD)
Description: TTPD is defined as time from the date of randomization to the first date of disease progression. For each participant who is not known to have had a progression of disease as of the data-inclusion cut-off date for a particular analysis, or who has died without progression of disease, TTPD will be censored for that analysis at the date of the participant's last tumor assessment prior to that cut-off date. TTPD was analyzed twice: (1) excluding clinical progressions of disease (that is,those not defined according to the RECIST version 1.1 criteria ), and (2) including clinical progressions. Progressive disease (PD) was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. Also, the sum must also demonstrate an absolute increase of at least 5 millimeter (mm). The appearance of one or more new lesions is also considered progression.
Time Frame: Randomization to Progressive Disease (Up To 58.78 Months)
Population: All participants who received at least 1 dose of study drug. Participants censored: Gefitinib/Pemetrexed =31, Gefitinib=4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 250 mg Gefitinib/500 mg Pemetrexed | 250 mg Gefitinib
Number analyzed (Participants) | 126 | 65
months | 16.23 [12.58 to 18.73] | 10.94 [9.66 to 13.83]
Statistical Analysis 1: Comparison: 250 mg Gefitinib/500 mg Pemetrexed vs 250 mg Gefitinib; Test type: Superiority or Other; p = 0.005, Regression, Cox — 1 sided; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.46 to 0.90]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to the date of death from any cause. Survival time is censored at the date of last contact for participants who are still alive or lost to follow up.
Time Frame: Randomization to Date of Death Due to Any Cause (Up To 67.12 Months)
Population: All participants who received at least 1 dose of study drug. Participants censored: Gefitinib/Pemetrexed =54, Gefitinib=26
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 250 mg Gefitinib/500 mg Pemetrexed | 250 mg Gefitinib
Number analyzed (Participants) | 126 | 65
Months | 43.43 [33.35 to 50.83] | 36.76 [26.74 to 42.64]
Statistical Analysis 1: Comparison: 250 mg Gefitinib/500 mg Pemetrexed vs 250 mg Gefitinib; Test type: Superiority or Other; p = 0.105, Regression, Cox — 1 sided; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.51 to 1.16]

4. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) (Overall Response Rate [ORR])
Description: ORR is the best response of complete response (CR) or partial response (PR) as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). Complete Response (CR) is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Tumor marker results must have normalized. Partial Response (PR) is defined at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters.
Time Frame: Randomization to Progressive Disease (Up to 57.36 Months)
Population: All participants who received at least 1 dose of study. Participants censored: Gefitinib/Pemetrexed =17, Gefitinib=3
Measure: Number; unit: percentage of participants
Arm/Group | 250 mg Gefitinib/500 mg Pemetrexed | 250 mg Gefitinib
Number analyzed (Participants) | 125 | 65
percentage of participants | 80.2 | 73.8

5. Secondary Outcome: Percentage of Participants With CR, PR, and Stable Disease (SD) (Disease Control Rate [DCR])
Description: Disease control rate is the percentage of participants with a confirmed CR, PR or SD as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST version 1.1) criteria. CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Tumor marker results must have normalized. PR is defined at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Randomization to Progressive Disease (Up To 57.36 Months)
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 250 mg Gefitinib/500 mg Pemetrexed | 250 mg Gefitinib
Number analyzed (Participants) | 125 | 65
percentage of participants | 92.9 | 93.8

6. Secondary Outcome: Duration of Response (DoR)
Description: DoR was defined as the time from the date of the first CR or PR to the first date of Progressive Disease (PD) ( RECIST 1.1 Criteria) or death from any cause.CR is the disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm.Tumor marker results must have normalized. PR is defined as at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters. PD was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. Also,the sum must also demonstrate an absolute increase of at least 5 mm.The appearance of one or more new lesions is also considered progression. Participants not known to have died or to have had progression of disease as of the data-inclusion cut-off date for a particular analysis,duration of tumor response was censored at the date of the participants last tumor assessment prior to that cut-off date.
Time Frame: First Observation of CR or PR to Progressive Disease or Death Due to Any Cause (Up To 57.36 Months)
Population: All randomized participants who received at least 1 dose of drug. Participants censored: Gefitinib/Pemetrexed =30, Gefitinib=7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 250 mg Gefitinib/500 mg Pemetrexed | 250 mg Gefitinib
Number analyzed (Participants) | 101 | 48
Months | 15.44 [10.87 to 17.71] | 11.30 [8.31 to 16.36]

7. Secondary Outcome: Time to Worsening of Symptom (TWS) as Per Lung Cancer Symptom Scale (LCSS)
Description: TWS was the elapsed time from the date of randomization to the first date of worsening in any one of the 6 LCSS symptoms. The LCSS (patient and observer) were administered at baseline and at the end of each 21-day cycle, until disease progression, and at short-term follow-up. Content for the patient version -collected using a visual analog scale (VAS) anchored at 0 and 100, respectively representing the best and worst outcome- included 6 disease-specific measures: (appetite, fatigue, cough, dyspnea, hemoptysis and pain) and 3 summary consequences of lung cancer (overall symptom burden, diminished normal activities, and lowered quality-of-life).The observer version included only the 6 disease-specific measures and the responses were collected using a 5-point ordinal scale that was reverse coded with 0 and 100 respectively representing the worst and best outcome.TWS was censored at the date of the last LCSS assessment for participants who were not known to have LCSS worsening.
Time Frame: Baseline to Progressive Disease (Up To 50 Months )
Population: Participants who received at least 1 dose of study drug & had evaluable events. Censored participants: a:52,32; b:60,32;c:68,43;d:73,39;e:97,43;f:78,45;g:64,38;h:54,37;i: 59,35; j:59,40;k:52,33;l:83,45;m:79,43;n:100,56;o:82,32 for 250 mg Gefitinib/500 mg Pemetrexed and 250 mg Gefitinib arms respectively.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 250 mg Gefitinib/500 mg Pemetrexed | 250 mg Gefitinib
Number analyzed (Participants) | 125 | 65
months
  a. Loss of Appetite (Patient-rated): number analyzed (Participants) | 73 | 33
  a. Loss of Appetite (Patient-rated) | 5.39 [3.68 to 12.29] | 7.66 [3.52 to NA] — There were insufficient events to support the statistical estimate of the 95% upper limit confidence interval.
  b. Fatigue (Patient-rated): number analyzed (Participants) | 65 | 33
  b. Fatigue (Patient-rated) | 8.51 [4.47 to 25.46] | 7.66 [2.79 to NA] — There were insufficient events to support the statistical estimate of the 95% upper limit confidence interval.
  c. Cough (Patient-rated): number analyzed (Participants) | 57 | 22
  c. Cough (Patient-rated) | 18.76 [8.15 to NA] — There were insufficient events to support the statistical estimate of the 95% upper limit confidence interval. | NA [11.79 to NA] — There were insufficient events to support the statistical estimate of the median and 95% upper limit confidence interval.
  d. Dyspnea (Patient-rated): number analyzed (Participants) | 52 | 26
  d. Dyspnea (Patient-rated) | 18.76 [11.66 to NA] — There were insufficient events to support the statistical estimate of the 95% upper limit confidence interval. | 24.87 [9.07 to NA] — There were insufficient events to support the statistical estimate of the 95% upper limit confidence interval.
  e. Hemoptysis (Patient-rated): number analyzed (Participants) | 28 | 22
  e. Hemoptysis (Patient-rated) | NA [21.06 to NA] — There were insufficient events to support the statistical estimate of the median and 95% upper limit confidence interval. | NA [10.68 to NA] — There were insufficient events to support the statistical estimate of the median and 95% upper limit confidence interval.
  f. Pain (Patient-rated): number analyzed (Participants) | 47 | 20
  f. Pain (Patient-rated) | 34.83 [16.03 to NA] — There were insufficient events to support the statistical estimate of the 95% upper limit confidence interval. | NA [15.47 to NA] — There were insufficient events to support the statistical estimate of the median and 95% upper limit confidence interval.
  g. Overall Symptoms (Patient-rated): number analyzed (Participants) | 61 | 27
  g. Overall Symptoms (Patient-rated) | 10.12 [5.85 to 21.55] | 30.46 [8.34 to NA] — There were insufficient events to support the statistical estimate of the 95% upper limit confidence interval.
  h. Interference (Patient-rated): number analyzed (Participants) | 71 | 28
  h. Interference (Patient-rated) | 5.72 [3.58 to 12.58] | 24.71 [9.72 to NA] — There were insufficient events to support the statistical estimate of the 95% upper limit confidence interval.
  i. Quality of Life (Patient-rated): number analyzed (Participants) | 66 | 30
  i. Quality of Life (Patient-rated) | 13.40 [4.24 to 34.83] | 10.61 [5.29 to NA] — There were insufficient events to support the statistical estimate of the 95% upper limit confidence interval.
  j. Loss of Appetite (Observer-rated): number analyzed (Participants) | 66 | 25
  j. Loss of Appetite (Observer-rated) | 8.61 [5.36 to 18.73] | 34.10 [11.14 to NA] — There were insufficient events to support the statistical estimate of the 95% upper limit confidence interval.
  k. Fatigue (Observer-rated): number analyzed (Participants) | 73 | 32
  k. Fatigue (Observer-rated) | 7.52 [5.09 to 13.93] | 12.98 [4.17 to NA] — There were insufficient events to support the statistical estimate of the 95% upper limit confidence interval.
  l. Cough (Observer-rated): number analyzed (Participants) | 42 | 20
  l. Cough (Observer-rated) | 41.92 [19.68 to NA] — There were insufficient events to support the statistical estimate of the 95% upper limit confidence interval. | NA [23.26 to NA] — There were insufficient events to support the statistical estimate of the median and 95% upper limit confidence interval.
  m. Dyspnea (Observer-rated): number analyzed (Participants) | 46 | 22
  m. Dyspnea (Observer-rated) | NA [15.31 to NA] — There were insufficient events to support the statistical estimate of the median and 95% upper limit confidence interval. | NA [19.32 to NA] — There were insufficient events to support the statistical estimate of the median and 95% upper limit confidence interval.
  n. Hemoptysis (Observer-rated): number analyzed (Participants) | 25 | 9
  n. Hemoptysis (Observer-rated) | NA [26.74 to NA] — There were insufficient events to support the statistical estimate of the median and 95% upper limit confidence interval. | NA [NA to NA] — There were insufficient events to support the statistical estimate of the median and 95% confidence interval.
  o. Pain (Observer-rated): number analyzed (Participants) | 43 | 33
  o. Pain (Observer-rated) | 34.83 [19.65 to NA] — There were insufficient events to support the statistical estimate of the 95% upper limit confidence interval. | 10.51 [4.90 to 35.88]
Statistical Analysis 1: Comparison: 250 mg Gefitinib/500 mg Pemetrexed vs 250 mg Gefitinib; Patient-rated Loss of Appetite: Time to worsening of symptom (TWS) was measured from the date of randomization to the first date of a 15-millimeter(mm) worsening from baseline on a scale of 0 (no symptoms) to 100 (as much as it could be); Test type: Superiority; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.77 to 1.78]
Statistical Analysis 2: Comparison: 250 mg Gefitinib/500 mg Pemetrexed vs 250 mg Gefitinib; Patient-rated Fatigue: Time to worsening of symptom (TWS) was measured from the date of randomization to the first date of a 15-millimeter(mm) worsening from baseline on a scale of 0 (no symptoms) to 100 (as much as it could be); Test type: Superiority; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.60 to 1.42]
Statistical Analysis 3: Comparison: 250 mg Gefitinib/500 mg Pemetrexed vs 250 mg Gefitinib; Patient-rated Cough: Time to worsening of symptom (TWS) was measured from the date of randomization to the first date of a 15-millimeter(mm) worsening from baseline on a scale of 0 (no symptoms) to 100 (as much as it could be); Test type: Superiority; Hazard Ratio (HR) = 1.39, 95% CI 2-sided [0.84 to 2.30]
Statistical Analysis 4: Comparison: 250 mg Gefitinib/500 mg Pemetrexed vs 250 mg Gefitinib; Patient-rated Dyspnea: Time to worsening of symptom (TWS) was measured from the date of randomization to the first date of a 15-millimeter(mm) worsening from baseline on a scale of 0 (no symptoms) to 100 (as much as it could be); Test type: Superiority; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.65 to 1.71]
Statistical Analysis 5: Comparison: 250 mg Gefitinib/500 mg Pemetrexed vs 250 mg Gefitinib; Patient-rated Hemoptysis: Time to worsening of symptom (TWS) was measured from the date of randomization to the first date of a 15-millimeter(mm) worsening from baseline on a scale of 0 (no symptoms) to 100 (as much as it could be); Test type: Superiority; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.32 to 1.02]
Statistical Analysis 6: Comparison: 250 mg Gefitinib/500 mg Pemetrexed vs 250 mg Gefitinib; Patient-rated Pain: Time to worsening of symptom (TWS) was measured from the date of randomization to the first date of a 15-millimeter(mm) worsening from baseline on a scale of 0 (no symptoms) to 100 (as much as it could be); Test type: Superiority; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.64 to 1.91]
Statistical Analysis 7: Comparison: 250 mg Gefitinib/500 mg Pemetrexed vs 250 mg Gefitinib; Patient-rated Overall Symptoms: Time to worsening of symptom (TWS) was measured from the date of randomization to the first date of a 15-millimeter(mm) worsening from baseline on a scale of 0 (no symptoms) to 100 (as much as it could be); Test type: Superiority; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.68 to 1.77]
Statistical Analysis 8: Comparison: 250 mg Gefitinib/500 mg Pemetrexed vs 250 mg Gefitinib; Patient-rated Interference: Time to worsening of symptom (TWS) was measured from the date of randomization to the first date of a 15-millimeter(mm) worsening from baseline on a scale of 0 (no symptoms) to 100 (as much as it could be); Test type: Superiority; Hazard Ratio (HR) = 1.38, 95% CI 2-sided [0.88 to 2.17]
Statistical Analysis 9: Comparison: 250 mg Gefitinib/500 mg Pemetrexed vs 250 mg Gefitinib; Patient-rated Quality of Life: Time to worsening of symptom (TWS) was measured from the date of randomization to the first date of a 15-millimeter(mm) worsening from baseline on a scale of 0 (no symptoms) to 100 (as much as it could be); Test type: Superiority; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.72 to 1.74]
Statistical Analysis 10: Comparison: 250 mg Gefitinib/500 mg Pemetrexed vs 250 mg Gefitinib; Observer-rated Loss of Appetite: Time to worsening of symptom (TWS) was measured from the date of randomization to the first date of a 15-millimeter(mm) worsening from baseline on a scale of 0 (Severe) to 100 (None). This scoring system is the reverse of the patient scale. The observer scale is a categorical 5-point scale and specific descriptors are provided with each questions for each of the scores (0,25,50,75 and 100); Test type: Superiority; Hazard Ratio (HR) = 1.56, 95% CI 2-sided [0.97 to 2.49]
Statistical Analysis 11: Comparison: 250 mg Gefitinib/500 mg Pemetrexed vs 250 mg Gefitinib; Observer-rated Fatigue: Time to worsening of symptom (TWS) was measured from the date of randomization to the first date of a 15-millimeter(mm) worsening from baseline on a scale of 0 (Severe) to 100 (None). This scoring system is the reverse of the patient scale. The observer scale is a categorical 5-point scale and specific descriptors are provided with each questions for each of the scores (0,25,50,75 and 100); Test type: Superiority; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [0.82 to 1.93]
Statistical Analysis 12: Comparison: 250 mg Gefitinib/500 mg Pemetrexed vs 250 mg Gefitinib; Observer-rated Cough:Time to worsening of symptom (TWS) was measured from the date of randomization to the first date of a 15-millimeter(mm) worsening from baseline on a scale of 0 (Severe) to 100 (None). This scoring system is the reverse of the patient scale. The observer scale is a categorical 5-point scale and specific descriptors are provided with each questions for each of the scores (0,25,50,75 and 100); Test type: Superiority; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.72 to 2.15]
Statistical Analysis 13: Comparison: 250 mg Gefitinib/500 mg Pemetrexed vs 250 mg Gefitinib; Observer-rated Dyspnea: Time to worsening of symptom (TWS) was measured from the date of randomization to the first date of a 15-millimeter(mm) worsening from baseline on a scale of 0 (Severe) to 100 (None). This scoring system is the reverse of the patient scale. The observer scale is a categorical 5-point scale and specific descriptors are provided with each questions for each of the scores (0,25,50,75 and 100); Test type: Superiority; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.64 to 1.83]
Statistical Analysis 14: Comparison: 250 mg Gefitinib/500 mg Pemetrexed vs 250 mg Gefitinib; Observer-rated Hemoptysis: Time to worsening of symptom (TWS) was measured from the date of randomization to the first date of a 15-millimeter(mm) worsening from baseline on a scale of 0 (Severe) to 100 (None). This scoring system is the reverse of the patient scale. The observer scale is a categorical 5-point scale and specific descriptors are provided with each questions for each of the scores (0,25,50,75 and 100); Test type: Superiority; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [0.60 to 2.91]
Statistical Analysis 15: Comparison: 250 mg Gefitinib/500 mg Pemetrexed vs 250 mg Gefitinib; Observer-rated Pain: Time to worsening of symptom (TWS) was measured from the date of randomization to the first date of a 15-millimeter(mm) worsening from baseline on a scale of 0 (Severe) to 100 (None). This scoring system is the reverse of the patient scale. The observer scale is a categorical 5-point scale and specific descriptors are provided with each questions for each of the scores (0,25,50,75 and 100); Test type: Superiority; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.41 to 1.03]

ADVERSE EVENTS:
Description: All participants who received at least 1 dose of study drug.
Arm/Group | 250 mg Gefitinib/500 mg Pemetrexed | 250 mg Gefitinib
Serious Adverse Events (participants affected / at risk) | 31/126 | 9/65
Other Adverse Events (participants affected / at risk) | 123/126 | 63/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 250 mg Gefitinib/500 mg Pemetrexed (N=126) | 250 mg Gefitinib (N=65)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 2 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 4 (4) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Biopsy lung (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary resection (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 250 mg Gefitinib/500 mg Pemetrexed (N=126) | 250 mg Gefitinib (N=65)
Anaemia (Blood and lymphatic system disorders) | 33 (41) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (5) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Corneal dystrophy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Cupulolithiasis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 2 (4)
Inner ear disorder (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 5 (10) | 2 (2)
Asthenopia (Eye disorders) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 8 (8) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 1 (1)
Conjunctival oedema (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 13 (15) | 1 (1)
Ectropion (Eye disorders) | 1 (1) | 0 (0)
Entropion (Eye disorders) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 4 (5) | 0 (0)
Eyelid oedema (Eye disorders) | 2 (3) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 13 (13) | 1 (1)
Myopia (Eye disorders) | 2 (2) | 0 (0)
Open angle glaucoma (Eye disorders) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 1 (1) | 0 (0)
Presbyopia (Eye disorders) | 2 (2) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Trichiasis (Eye disorders) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 8 (8) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 10 (12) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 9 (10) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 6 (8) | 2 (3)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 28 (37) | 8 (9)
Dental caries (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 69 (132) | 35 (62)
Dry mouth (Gastrointestinal disorders) | 6 (8) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 8 (10) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (4) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 6 (6) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 (12) | 4 (6)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (2)
Haemorrhoids (Gastrointestinal disorders) | 5 (6) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 4 (4) | 3 (5)
Nausea (Gastrointestinal disorders) | 41 (88) | 9 (11)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oral pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 5 (5) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 47 (86) | 15 (29)
Tooth loss (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 7 (9) | 1 (1)
Vomiting (Gastrointestinal disorders) | 24 (40) | 6 (9)
Asthenia (General disorders) | 4 (4) | 3 (3)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 4 (4) | 1 (1)
Chest pain (General disorders) | 4 (4) | 3 (3)
Chills (General disorders) | 2 (3) | 1 (1)
Face oedema (General disorders) | 17 (19) | 3 (3)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 45 (77) | 15 (17)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Granuloma (General disorders) | 0 (0) | 1 (1)
Induration (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 9 (11) | 3 (4)
Malaise (General disorders) | 13 (15) | 6 (7)
Mucosal erosion (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 12 (17) | 2 (2)
Oedema peripheral (General disorders) | 23 (48) | 1 (1)
Pain (General disorders) | 2 (2) | 2 (2)
Peripheral swelling (General disorders) | 2 (3) | 1 (1)
Pyrexia (General disorders) | 15 (18) | 5 (7)
Sluggishness (General disorders) | 1 (1) | 0 (0)
Soft tissue inflammation (General disorders) | 0 (0) | 1 (1)
Xerosis (General disorders) | 6 (6) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (3) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 2 (3) | 1 (1)
Amyloidosis (Immune system disorders) | 0 (0) | 1 (1)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (2)
Angular cheilitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 7 (8) | 1 (3)
Conjunctivitis (Infections and infestations) | 10 (13) | 3 (3)
Cystitis (Infections and infestations) | 5 (6) | 1 (2)
Dermatophytosis of nail (Infections and infestations) | 1 (1) | 1 (1)
Eye infection (Infections and infestations) | 3 (3) | 0 (0)
Folliculitis (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gingival abscess (Infections and infestations) | 1 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 3 (3) | 1 (1)
Herpes zoster infection neurological (Infections and infestations) | 1 (2) | 0 (0)
Infection (Infections and infestations) | 2 (8) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 4 (4) | 2 (2)
Localised infection (Infections and infestations) | 0 (0) | 1 (2)
Lung infection (Infections and infestations) | 5 (5) | 2 (2)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Otitis media (Infections and infestations) | 2 (2) | 1 (1)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 40 (53) | 14 (20)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 3 (4)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyuria (Infections and infestations) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 11 (16) | 5 (5)
Rhinitis (Infections and infestations) | 5 (5) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 5 (5) | 2 (2)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 5 (5) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1)
Tracheitis (Infections and infestations) | 2 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 17 (28) | 6 (17)
Urinary tract infection (Infections and infestations) | 8 (9) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Viral hepatitis carrier (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvitis (Infections and infestations) | 2/82 (2) | 0/41 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dental restoration failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Fractured coccyx (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 52 (72) | 25 (41)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 57 (83) | 24 (35)
Blood alkaline phosphatase increased (Investigations) | 10 (14) | 5 (5)
Blood bilirubin increased (Investigations) | 4 (7) | 10 (20)
Blood cholesterol increased (Investigations) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 11 (15) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 1 (1)
Blood urea increased (Investigations) | 1 (1) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Computerised tomogram thorax abnormal (Investigations) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 7 (26) | 0 (0)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 10 (14) | 2 (2)
Haemoglobin decreased (Investigations) | 2 (2) | 2 (3)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 3 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 6 (7) | 0 (0)
Monocyte count increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 26 (66) | 2 (3)
Neutrophil count increased (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 6 (8) | 3 (3)
Platelet count increased (Investigations) | 1 (2) | 0 (0)
Total bile acids increased (Investigations) | 1 (1) | 4 (6)
Weight decreased (Investigations) | 24 (30) | 8 (10)
Weight increased (Investigations) | 7 (12) | 0 (0)
White blood cell count decreased (Investigations) | 24 (60) | 7 (15)
White blood cell count increased (Investigations) | 3 (6) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 49 (96) | 17 (20)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 11 (14) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (6) | 3 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (11) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (5) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 7 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 4 (4)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oral neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 1 (1)
Clumsiness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 21 (26) | 8 (12)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 17 (17) | 4 (4)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 14 (17) | 8 (12)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 2 (2)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (4) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (9) | 3 (3)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 2 (3) | 1 (1)
Tremor (Nervous system disorders) | 3 (4) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Vascular dementia (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (4) | 3 (3)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 23 (29) | 6 (8)
Persistent depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 3 (3) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 4 (4) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 3 (3) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 3 (3) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1/82 (1) | 0/41 (0)
Pelvic haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Pruritus genital (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1/82 (1) | 0/41 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1/82 (1) | 0/41 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/82 (1) | 0/41 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (41) | 11 (18)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (20) | 9 (11)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (6) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 7 (8)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 (22) | 6 (6)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (11) | 6 (6)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tracheal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Vocal cord inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (12) | 3 (3)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 49 (69) | 29 (37)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 33 (37) | 24 (30)
Eczema (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 44 (58) | 22 (32)
Rash (Skin and subcutaneous tissue disorders) | 21 (27) | 12 (15)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 19 (21) | 5 (5)
Rosacea (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 8 (10) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 16 (16) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Intraocular lens implant (Surgical and medical procedures) | 1 (1) | 0 (0)
Pericardial drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 8 (8) | 4 (4)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Internal haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days